CLINICAL TRIAL: NCT00546546
Title: Effect of Early Prescription of Immunosuppressants on First Three-year Course of Crohn's Disease
Brief Title: Early Immunosuppressants in Crohn's Disease
Acronym: RAPID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2004-2
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2011-08

CONDITIONS: Crohn's Disease
Keywords: Crohn; immunosuppressants; natural history; steroids
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control = conventional treatment (No Intervention): conventional treatment: use of immunosuppressants only if steroid dependency or chronic active disease
- Immunossuppresive treatment (Experimental): Switch to different immunosuppresive treatment in case of relapse.
  Interventions: Drug: early immunosuppressants (azathioprine, methotrexate)

INTERVENTIONS:
Drug: early immunosuppressants (azathioprine, methotrexate) — azathioprine 2.5 mg/kg/day SC methotrexate 25 mg/week if aza not tolerated
  Other Names: Azathioprine = brand name = Imurel
  Arms: Immunossuppresive treatment

SUMMARY:
Pluricentric randomized study comparing two therapeutic strategies at beginning of Crohn's disease: early immunosuppressants (prescription within the six first months following diagnosis) vs. conventional strategy (immunosuppressants given only in case of steroid failure, in a selected group of patients being at high risk of disabling course. The hypothesis is that immunosuppressants given early may improve the disease course during the 3 following years in this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* > 18 yr old
* diagnosis of Crohn's disease
* intestinal lesions demonstrated during the last 6 months
* disease duration < 6 months
* patients at high risk of disabling disease (having 2 criteria out of the 3 following: age < 40, perinanal disease, steroid for the first flare)

Exclusion Criteria:

* prior prescription of immunosuppressants
* severe course requiring early immunosuppressants (steroid resistance, xtensive disease, disabling perianal disease)
* intestinal resection
* active infectious disease including HIV
* hepatic failure
* renal failure
* pregnancy
* high probability of poor compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
number of 3-months periods with remission | 3 yrs

SECONDARY OUTCOMES:
3-yr cumulative steroid dose | 3 years
quality of life questionnaire | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Marc LEMANN, PhD, Study Director — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Jacques COSNES, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (26):
- France (26):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - CHU CAEN, Caen
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourrier, Colombes
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Chru Lille, Lille
  - Chu Marseille - Hopital Nord, Marseille
  - Ch Le Raincy Montfermeil, Montfermeil
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Georges Pompidou, Paris
  - Hopital Bichat, Paris
  - Institut Mutualiste Montsouris (Imm), Paris
  - Hopital Haut Leveque, Pessac
  - CHU LYON, Pierre-Bénite
  - Chu Reims, Reims
  - Chu Rouen, Rouen
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- [Background] Beaugerie L, Seksik P, Nion-Larmurier I, Gendre JP, Cosnes J. Predictors of Crohn's disease. Gastroenterology. 2006 Mar;130(3):650-6. doi: 10.1053/j.gastro.2005.12.019. PMID 16530505
- [Background] Cosnes J, Nion-Larmurier I, Beaugerie L, Afchain P, Tiret E, Gendre JP. Impact of the increasing use of immunosuppressants in Crohn's disease on the need for intestinal surgery. Gut. 2005 Feb;54(2):237-41. doi: 10.1136/gut.2004.045294. PMID 15647188
- [Derived] Cosnes J, Bourrier A, Laharie D, Nahon S, Bouhnik Y, Carbonnel F, Allez M, Dupas JL, Reimund JM, Savoye G, Jouet P, Moreau J, Mary JY, Colombel JF; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif (GETAID). Early administration of azathioprine vs conventional management of Crohn's Disease: a randomized controlled trial. Gastroenterology. 2013 Oct;145(4):758-65.e2; quiz e14-5. doi: 10.1053/j.gastro.2013.04.048. Epub 2013 Apr 30. PMID 23644079